CLINICAL TRIAL: NCT06843694
Title: Effect of Video Game Training on Student Nurses' Intervention in Adult Airway Obstruction: a Mixed Methods Study
Brief Title: Video Game Training on Intervention in Adult Airway Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Di̇lek Soylu, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024/02
Record Dates: First submitted 2025-01-18; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Airway Obstruction
Keywords: Airway obstruction; Video game; Nurse; Education
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Intervention Model Description: A pre-test-post-test control group and repeated-measures experimental design type
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researcher (3) was not involved in any stage of the training. He made the students practice on the mannequin without knowing their groups and collected the data. In this direction, a single blind technique was used. The interview for the qualitative data was conducted by the researcher (2) and he collected the qualitative study data as audio recordings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video Game (Experimental): The students in the video game group will be given training. The students in this group (n=30) will be divided into 4 groups and there will be 5 students in each group. The students will be given training about the Video Game (Lifesaver) by the researcher beforehand. The Video Game (Lifesaver-Cankurtaran); is a free video game developed by the Resuscitation Council in English. It can be downloaded for free from the Google Play Store on a computer, phone or tablet.
  Interventions: Other: video game
- Control group (No Intervention): A pre-test will be administered to each participant to test their knowledge of providing care to an adult with airway obstruction. A researcher who is blind to the student group will distribute the pre-test questionnaires (Personal Information Form, Adult Airway Obstruction Prevention and Management Information Form, Adult Airway Obstruction Prevention and Management Skills Form) to the participants and ensure that they are filled out. One week after the pre-test, both groups will be trained in a first and emergency aid course on the same day. The content of the training will be the same for both groups. The researcher (1) will provide a total of 90 minutes of training in the form of theoretical and classroom skills training. The researcher (2) will explain to the students in the intervention group how to download and use the video game. The control group will attend the course only once before the post-test.

INTERVENTIONS:
Other: video game — The students in the video game group will be given training. The students in this group (n=30) will be divided into 4 groups and each group will have 5 students. The students will be given training about the Video Game (Lifesaver) by the researcher beforehand. The Video Game (Lifesaver-Cankurtaran); is a free video game developed by the Resuscitation Council in English.
  Arms: Video Game

SUMMARY:
Foreign body aspiration occurs as a result of partial or complete airway obstruction. In the case of complete obstruction, mechanical asphyxia can lead to insufficient ventilation and oxygenation, leading to death. Basic life support education is generally provided in schools in Turkey using traditional education methods. First aid is one of the important professional skills that nurses need. Due to the crowded classroom environment, not all students can clearly see the skill applications performed by the instructors, and the applications can be interrupted by the students. The World Health Organization recommends mobile-based education applications as a comprehensive education method for health systems. The aim of this study is to compare the effects of Video Game and Classical Education methods in Adult Airway Obstruction education given to nursing students in a pre-test-post-test control group and repeated measures experimental design type. No international or national research was found on the subject. Therefore, the study is original. The research is a mixed-methods research with an embedded design model. The reason for choosing this type is that presenting qualitative and quantitative methods together allows researchers to see different perspectives and to reveal the relationships between the complex layers of the research questions in a clearer and more understandable way. The quantitative phase was conducted as a randomized controlled experimental design, while the qualitative phase was conducted using a simultaneous embedded design in the phenomenological design. The "Mixed Methods Research Methodology Development Checklist" was used as a guide in reporting this research. The sample size was calculated as 60. In data collection, information on socio-demographic characteristics will be collected with the "Introductory information form, semi-structured questionnaire form, Adult Airway Obstruction Prevention and Management Information Form and Adult Airway Obstruction Prevention and Management Skills Form". The surveys will be applied to the adults participating in the study through face-to-face interviews. Semi-structured questions will also be asked to 20-25 volunteers from different age groups and genders participating in the survey. Content analysis was used in the analysis of the qualitative data. Semi-structured questions were directed to students using a face-to-face interview technique and their answers were recorded with a voice recorder. The voice recordings were listened to repeatedly by the researchers and deciphered. After deciphering, qualitative analysis was performed with the code-category-thematic analysis process. Methodologically, inductive coding was followed in the analysis of the data. Max Qualitative Data Analysis (MAXQDA) Analytics Pro2024 program was used in the analysis.

Rigor and reflexivity Triangulation and verification; Qualitative analysis was performed by the second author, the other two authors examined all stages of the analysis to achieve the highest data quality and tested and approved the analysis according to the accuracy of each other's notes. This stage ensured the reliability of the analysis and verified the coding of the data. With this method, the reliability of the research, the meticulousness, credibility, reliability, transferability and appropriateness of the collected data were tested.

In quantitative data; The data belonging to the participants in the study were analyzed using SPSS Statistics 20.0. Descriptive statistics (n, %) were given for categorical variables. Compliance with normal distribution was assessed with the "Kolmogrov-Smirnov test". In order to test whether the scores obtained from two unrelated samples of quantitative variables differed significantly from each other, the "independent sample t test" was applied for parametric testing. In the analysis of the data, "Chi-square analysis" was performed to see the differences of qualitative data according to groups. "Pearson correlation test" was applied to evaluate the relationship between knowledge and skill level scores. "Reliability Analysis" was performed to test the reliability of the scales.

ELIGIBILITY:
Inclusion Criteria:

* Being an undergraduate student,
* Having taken an Internal Medicine and Surgical Nursing course,
* Not having previously received Adult Airway Obstruction Prevention and Management training,
* Not having any previous experience with video game-based learning in healthcare and not having problems with internet access.

Exclusion Criteria:

* Students who did not agree to participate in the study,
* Students who did not meet the inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Adult Airway Obstruction Prevention and Management Information Form | 1 hour and 1 month
  Adult Airway Obstruction Prevention and Management Information Form: The tool used to assess students' knowledge on preventing and managing adult airway obstruction was developed by researchers based on the American Heart Association (AHA) guidelines for providing emergency care to adults (2011) and the Republic of Turkey Ministry of Health standards (2021). It consists of 10 multiple-choice questions created to assess the knowledge level of students in both groups. Each question consists of 4 options, and each correct answer given by the researchers is calculated as "1" point, while incorrect or "I have no idea" answers are calculated as "0" points. The maximum score in this form is "10", while the minimum score is "0".

SECONDARY OUTCOMES:
Adult Airway Obstruction Prevention and Management Skill Form | 1 hour and 1 month
  Adult Airway Obstruction Prevention and Management Skill Form: The tool used to assess student skills in dealing with adult airway obstruction was developed by the study authors and was also based on the American Heart Association (AHA) guidelines for providing emergency care to adults (2011) and the Republic of Turkey Ministry of Health standards (2021) guidelines for providing emergency care to adults. The skill form consists of 30 actions; 1 for danger control, 1 for determining the type of obstruction, 1 for partial obstruction, 1 for complete obstruction, and 26 for intervention in people with complete obstruction. Students were assessed in 3 actions. These were:
  1. Adequate: "Students should be able to express and perform the TYD steps in order, completely and accurately."
  2. Needs improvement: "Students should be able to express and perform at least half of the TYD steps in order, completely and accurately."
  3. Inadequate: "Students expressing more than half of the TYD steps i

CONTACTS AND LOCATIONS:
Locations (1):
- Afsin Health College, Afşin, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller GE. The assessment of clinical skills/competence/performance. Acad Med. 1990 Sep;65(9 Suppl):S63-7. doi: 10.1097/00001888-199009000-00045. No abstract available. PMID 2400509
- [Background] Chen PJ, Liou WK. The effects of an augmented reality application developed for paediatric first aid training on the knowledge and skill levels of nursing students: An experimental controlled study. Nurse Educ Today. 2023 Jan;120:105629. doi: 10.1016/j.nedt.2022.105629. Epub 2022 Nov 8. PMID 36375385
- [Background] Chen PJ, Liou WK. Development and Application of AR-Based Assessment System for Infant Airway Obstruction First Aid Training. Children (Basel). 2022 Oct 26;9(11):1622. doi: 10.3390/children9111622. PMID 36360350
- [Background] Behboudi F, Pouralizadeh M, Yeganeh MR, Roushan ZA. The effect of education using a mobile application on knowledge and decision of Iranian mothers about prevention of foreign body aspiration and to relieve choking in children: A quasi-experimental study. J Pediatr Nurs. 2022 Jan-Feb;62:e77-e83. doi: 10.1016/j.pedn.2021.07.007. Epub 2021 Jul 30. PMID 34334255
- [Background] Kim SJ, Shin H, Lee J, Kang S, Bartlett R. A smartphone application to educate undergraduate nursing students about providing care for infant airway obstruction. Nurse Educ Today. 2017 Jan;48:145-152. doi: 10.1016/j.nedt.2016.10.006. Epub 2016 Oct 25. PMID 27810633